CLINICAL TRIAL: NCT05845359
Title: Randomized Control Study on the Effectiveness of Intraoperative Methadone on Postoperative Pain Control
Brief Title: Intraoperative Methadone for Postoperative Pain Control
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: IRB approval never received
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-14040
Record Dates: First submitted 2022-10-26; First posted 2023-05-06 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Bariatric Surgery Candidate
Keywords: methadone; bariatric surgery; pain management
MeSH Terms: conditions — Agnosia | interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methadone group (Experimental): Patients in this group will receive intraoperative methadone.
  Interventions: Drug: Methadone
- Control group (No Intervention): Patients in this group will receive saline (placebo), instead of methadone

INTERVENTIONS:
Drug: Methadone — One group will receive 10mg of methadone upon induction, while the other will receive a saline solution as placebo. We will see the effectiveness of methadone on postoperative pain management, while monitoring for opioid-related side effects.
  Arms: Methadone group

SUMMARY:
To compare patient pain perception and satisfaction as well as opioid-related side effects during inpatient and outpatient care when undergoing bariatric enhanced recovery after surgery protocols with and without methadone.

ELIGIBILITY:
Inclusion Criteria:

• All patients undergoing initial gastric sleeve resection

Exclusion Criteria:

* Age <18 years or >60 years
* Patients with BMI >60
* AHI > 30 (AHI = Apnea-Hypopnea Index), indicative of severe Obstructive Sleep Apnea (OSA)
* ASA IV or V (American Society of Anesthesiology physical status classification system)
* Patients taking opioids for chronic conditions in the last 10 days preceding the surgery
* Patients currently being treated for chronic opioid addiction
* Patients with severe psychiatric diagnoses
* Allergies to medications used in protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative opioid use | 24 hours postoperatively
  Postoperative opioid use will be determined by the amount of morphine consumed (milligram morphine equivalents, MME) at 24 hours postoperatively

SECONDARY OUTCOMES:
Total Postoperative opioid use | 48 hours postoperatively and approximately at 2 weeks (follow up visit upon discharge)
  Total postoperative opioid use will be determined by the total amount of morphine consumed (milligram morphine equivalents, MME) at 48 hours postoperatively and during follow up visit
Respiratory interventions | Up to 4 hours postoperatively
  The number of respiratory interventions required postoperatively per patient in the PACU (Post-anesthesia care unit) will be determined
Duration of hospital stay | Approximately 5 days postoperatively
  The average duration of hospitalization will be determined per patient
Patients Perception of Pain Management | 24 hours postoperatively
  Patients perceptions of pain management will be measured by administration of the International Pain Outcomes (IPO) questionnaire on Post-Operative Day 1 (POD 1). IPO will be used to assess key patient level outcomes of postoperative pain management and consists of 13 questions evaluating four outcome domains: 1) intensity of pain rated on Numeric Rating Scale (NRS) score (0 = no pain, 10 = worst possible pain); 2) interference of pain with activities and emotional well-being as determined by a score analogous to the NRS 0-10 scale above; 3) side effects of pain treatment, including nausea, drowsiness, itching, and dizziness, as determined by the NRS score >0; and 4) perception of care, treatment satisfaction and involvement in pain treatment decision-making on a scale from 0-10. Scores are aggregated per patient with higher overall scores indicative of a worsening perception of pain management.
Patients Perception of Pain Management | 2 days postoperatively
  Patients perceptions of pain management will be measured by administration of the International Pain Outcomes (IPO) questionnaire on POD 1 (Post-Operative Day 1). IPO will be used to assess key patient level outcomes of postoperative pain management and consists of 13 questions evaluating four outcome domains: 1) intensity of pain rated on numeric rating score (0 = no pain, 10 = worst possible pain); 2) interference of pain with activities and emotional well-being as determined by a score analogous to the 0-10 scale above; 3) side effects of pain treatment, including nausea, drowsiness, itching, and dizziness, as determined by the NRS score >0; and 4) perception of care, treatment satisfaction and involvement in pain treatment decision-making on a scale from 0-10. Scores are aggregated per patient with higher overall scores indicative of a worsening perception of pain management.
Sedation Score (POSS) | 2 days postoperatively
  Sedation score will be determined using the Pasero Opioid-induced Sedation Scale (POSS) in the Post-anesthesia Care Unit (PACU) and on the floor. Average scores will be tabulated per patient using a four point numeric rating scale. Scoring is as follows: 1 = Awake and alert; 2 = Slightly drowsy, easily aroused; 3 = Frequently drowsy, arousable, drifts off to sleep during conversation; 4 = Somnolent, minimal or no response to verbal and physical stimulation
Agitation and Sedation Severity (RASS) | 2 days postoperatively
  Agitation and Sedation severity will determined using the Richmond Agitation-Sedation Scale (RASS) in the PACU and on the floor. Average scores will be determined per patient using a numeric rating scale ranging from +4 to -5 where +4 = combative, +3 = very agitated, +2 = agitated, +1 = restless, 0 = alert and calm, -1: = drowsy, -2 = light sedation, -3 = moderate sedation, -4 = deep sedation, and -5 = unarousable. Ideal RASS scores range from -1 to 1.
Opioid-related side effects | Up to 2 days postoperatively
  Opioid related side effects including nausea, vomiting, pruritis, urinary retention, and necessity of supplemental oxygen will be recorded
Early Mobilization | Up to 2 days postoperatively
  The average duration of time to first ambulation after surgery will be recorded per patient
GI recovery time | Up to 2 days postoperatively
  The average duration of time to return of bowel function will be determined per patient
Adverse events due to procedure or anesthesia | Up to 2 days postoperatively
  Procedure related adverse events or adverse events related to anesthesia will be recorded
Pain Scores | After 30 minutes in the PACU; upon discharge from PACU (variable timepoint); at 6, 12, 18, and 24 hours after being on the in-patient floor; and at hospital discharge
  Pain scores will be assessed by a research assistant blinded to the study group at regular intervals. Numerical pain scores (0=no pain, 10=most pain) will be assigned on an 11 point scale ranging from 0 (no pain) to 10 (most pain). Since most patients who get bariatric surgery are discharged at POD 1, the research assistant will call the patient the morning of POD 2 to assess the pain score if not on the inpatient floor. If the patients are not yet discharged, the pain score will be assessed the morning of POD 2, otherwise pain scores will be collected as detailed in the time frame below.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Choi, MD, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: No